CLINICAL TRIAL: NCT05981547
Title: Insights Into Glucose Variability Using Continuous Glucose Monitoring in Mothers With Gestational Diabetes Compared to Mothers at High Risk of Gestational Diabetes Who Have a Negative Oral Glucose Tolerance Test.
Brief Title: Patterns and Glycaemic Endpoints for Diagnosing Gestational Diabetes
Acronym: PAGED-GDM
Status: Active, not recruiting | Type: Observational
Sponsor: Portsmouth Hospitals NHS Trust (Other Government)
Collaborators: Abbott (Industry)
Responsible Party: Sponsor
Other Study IDs: 325114
Record Dates: First submitted 2023-07-17; First posted 2023-08-08 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Gestational Diabetes
Keywords: GDM - gestational diabetes; CGM - continuous glucose monitoring; AGP - ambulatory glucose profile; OGTT - Oral glucose tolerance test; NICE - national institute for health and care excellence; JDANC - Joint diabetes antenatal clinic
MeSH Terms: conditions — Diabetes, Gestational

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Device: Libre 3 continuous glucose monitoring sensor — Libre 3 CGM sensor applied to women prior to their Oral Glucose Tolerance test.

SUMMARY:
Gestational diabetes (GDM) develops during pregnancy and is becoming increasingly common. The condition is associated with adverse outcomes for mother and baby during both the pregnancy and delivery period. This study compares glucose variability (recorded by a continuous glucose monitoring (CGM) sensor) in pregnant women who have been diagnosed with GDM with pregnant woman who do not have the diagnosis but are at high risk. The sensors will be applied to 400 participants around the time of their standard test for GDM, with a randomly selected 60 of these patients forming a sub-group later in the study to assess for progression of high blood glucose. At present, a positive oral glucose tolerance test (OGTT) is used to confirm the diagnosis of GDM but the test can be unreliable leading to potential diagnostic error. CGM devices are used extensively in the management of Type 1 diabetes and GDM, and have also shown potential to be used in the diagnosis of Type 2 diabetes.

If this study can demonstrate similar trends in glucose variability between OGTT positive patients and those who are OGTT negative but are at high risk for the condition, then further research into the utility of CGM as a diagnostic alternative or supplement to the OGTT would be indicated.

The investigators will recruit 400 patients at high risk for GDM, give them a blinded CGM device, and compare the CGM glucose data with their OGTT result, their initial risk factors for GDM, their pregnancy outcome and their need for treatment. The investigators will use the data to test our hypothesis that a positive OGTT result does not predict hyperglycaemia in pregnancy.

DETAILED DESCRIPTION:
Gestational Diabetes (GDM) is associated with higher than normal blood sugar levels in pregnant women which has the potential to harm the baby and mother. The condition resolves with delivery of the baby, but during the pregnancy there is a limited time window for diagnosis and treatment before harm may be caused.

GDM is thought to affect up to 32% of pregnancies and is becoming more common due to rising rates of obesity and maternal age. The current recommended practice in the UK for the diagnosis of GDM is to use the oral glucose tolerance test (OGTT), which is two plasma blood glucose tests (one at baseline and one 2 hours after a glucose load) performed on expectant mothers who have at least one risk factor for GDM at 28 weeks gestation. This method is not standard internationally, with some countries using the test on all woman who fall pregnant, others adhering to different diagnostic thresholds, and others performing the test in a different way. Furthermore, there is no international consensus on the best way to diagnoses GDM. The challenge in diagnosing the condition arises because the results of the OGTT relies upon only two glucose measurements and therefore are not always accurate, meaning that some expectant mothers with GDM are missed, and others who do not have GDM are incorrectly told they have the condition.

Pregnant women who develop GDM but are not identified by the OGTT may suffer complications which could have been avoided with glucose lowering therapy, whilst woman who are incorrectly diagnosed with the condition may have their pregnancies unnecessarily medicalised, both of which places extra burden on the healthcare system. Therefore, improving the accuracy of the diagnosis of GDM has the potential to improve outcomes in pregnancies worldwide (and significantly impact upon current practice).

Recent technological advances in the field of diabetes care have seen the emergence of continuous glucose monitoring (CGM) - digital sensors placed on a patient's skin which constantly read the blood sugar level and communicate with their smart phone. Data from the CGM sensor is sent via Bluetooth to the smart phone, and using software downloaded in an app, is converted into a graphical summary illustration called an 'ambulatory glucose profile' (AGP) allowing for better treatment decisions to be made.

CGM devices are revolutionising the monitoring and treatment of diabetes, including GDM, however they are not utilised for diagnostic purposes. This study examines the challenging task of accurately diagnosing GDM by comparing the CGM data of patients with GDM with the CGM data of individuals at high risk of GDM (who are OGTT negative) to determine if the OGTT result is predictive of high blood glucose.

The glucose data from CGM devices in woman who test positive on the OGTT will be compared with women who are high risk for GDM but test negative, whilst also correlating with pregnancy outcomes such as need for treatment or complications. The study aims to test the hypothesis that a positive OGTT may not predict hyperglycaemia in pregnancy. If the hypothesis is proven correct, it may suggest that CGM/AGP has the potential to improve the current methodology of testing for GDM and that further studies examining this would be recommended.

The study will be undertaken in the Academic department of Diabetes and Endocrinology and the Joint diabetes antenatal clinic at Queen Alexandra Hospital, Portsmouth Hospitals University NHS trust. Participants will be pregnant women who have been identified according to established NICE criteria as being suitable for screening for GDM. Woman with any of the following risk factors are offered a screening test (OGTT) for GDM as per standard NHS care: BMI above 30kg/m², previous macrosomic baby weighing 4.5kg or more, previous GDM, family history of diabetes (first-degree relative with diabetes), an ethnicity with a high prevalence of diabetes. Patients with the risk factor 'previous GDM' will be excluded from the study as this prior diagnosis may influence behaviour in the current pregnancy. The risk assessment is undertaken during their booking appointment at 12 weeks gestation.

Participants will be identified using the hospital's electronic maternity records system, contacted at the earliest opportunity and given the participant information sheet (PIS). Patients will be given sufficient time to read the PIS (at least 24 hours) after which eligibility criteria will be checked and informed consent taken. This will take place during 12-26 weeks gestation. All participants will continue to receive antenatal care. The investigators will recruit 400 participants onto the study.

Study visit 1: (26-27 weeks gestation) This will be an in person visit at our site which is in addition to standard antenatal care. This is the only visit that is additional to standard NHS care for the majority of the study cohort. The study process will be discussed in full and any questions answered. A CGM device (freestyle Libre sensor) will be applied to the patient. It collects data automatically and is blinded.

Study visit 2: (28 weeks Gestation - OGTT date) When the participants attend for their OGTT they will have further opportunity to interact with the study team (all of whom are involved in the routine delivery of NHS maternity diabetes care) and any issues will be addressed. Their CGM devices will be removed at the end of the data capture period. The data from their OGTT test will be compared with their CGM data.

Sub-Group Study visit 3: 32 weeks gestation Of the 400 patients, 60 will be randomly selected (to include 30 OGTT positive and 30 OGTT negative patients) to form a sub-group. Patients in this sub-group will be invited prior to their standard NHS 32 week maternity visit to receive a further CGM device which will be applied on the day of the visit. The sub-group analysis is to assess for progression of glycaemia in both OGTT positive and negative groups.

Further study visits (up until end of gestation) Participants who tested positive on their OGTT are diagnosed with GDM and are usually followed up fortnightly in the JDANC clinic as part of routine NHS care. The study team will use information from these visits to inform the previously stated secondary objectives.

Follow up:

Patients will not be required to fill in questionnaires or attend further study visits in the follow up period. Electronic data will be collected on birth outcome; including mode of delivery, birth weight, premature delivery, any adverse fetal outcomes or neonatal hypoglycaemia. Data will be collected on the participants' 3 month post-partum HbA1c test that assess for resolution of GDM. This is a routine test that will not be undertaken by the study team but will be easily accessible on the electronic hospital record.

ELIGIBILITY:
Inclusion Criteria:

* Female aged 18 years of above
* Between 12-26 weeks gestation
* Identified by NICE as having one or more independent risk factor for GDM
* Suitable for the standard care pathway under the joint antenatal clinic for GDM
* Willing and able to give informed consent.

Exclusion Criteria:

* Pre-existing diabetes
* Previous GDM
* Unsuitable for standard joint antenatal clinic pathway
* Known allergy to freestyle libre adhesive pad
* Planning to move geographical area during the study timeframe
* Participating in a different study that could interfere with glucose levels or affect ability to participate.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Needs to be female aged 18 or above, between 12-26 weeks gestation.
Study Population: The investigators will recruit 400 patients, with the expectation that approximately 120 of these will have confirmed GDM following an OGTT. Of these patients, we expect 50% will require glucose lowering therapy (metformin and/or insulin) and 50% willo manage their GDM with dietary measures. The sample sizes are derived from the fact that CGM (AGP) comparisons across groups require n=18-20 in each group to give 80% power to detect clinically significant differences and so our sample size calculations are driven by making sure no sub-group has less than 20 subjects in it. The total of 120 positive OGTTs can be further sub-divided by how they achieved the positive OGTT (fasting, post glucose load, or both).
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2023-11-22 (Actual); Primary Completion 2026-06-21 (Estimated); Study Completion 2026-06-21 (Estimated)

PRIMARY OUTCOMES:
Time in range on CGM data (glucose 3.9-10) | 12 months
  Assessed glucose parameters and trends on ambulatory glucose profile provided by continuous glucose monitoring data.
Time in hyperglycaemia (glucose >10) | 12 months
  Assessed glucose parameters and trends on ambulatory glucose profile provided by continuous glucose monitoring data.
Glucose management indicator (GMI) - 'estimated A1c' | 12 months
  CGM device 'estimated A1c' calculation from the available data. This correlates with average glucose level
Glucose variability | 12 months
  Measure provided by CGM device referring to the amplitude and frequency of variation from the average glucose level. This does not directly correlate with average glucose level.

SECONDARY OUTCOMES:
Glucose lowering therapy. | 12 months
  Whether metformin and/or insulin was initiated and requirement for dose adjustment
A analysis of CGM glucose data for progression of glycaemia in a sub group | 12 months
  60 of the 400 patients will be offered a further CGM device to assess for progression of glycaemia a further 4-6 weeks into their pregnancy from the initial sensor fitting/glucose capture period. For example <10% would be low glucose variability (non-diabetic population), whereas >40% would be significant glucose variability.

CONTACTS AND LOCATIONS:
Overall Officials: Laura Marshall, Bsc, Study Chair — Portsmouth Hospitals University NHS Trust
Locations (1):
- Portsmouth Hospitals University NHS Trust, Portsmouth, United Kingdom

IPD SHARING:
Plan to Share IPD: No
IPD will not be available to other researchers